CLINICAL TRIAL: NCT00124501
Title: The Impact of Biofeedback-Assisted Relaxation Training on Pain and Functional Disability in Children Diagnosed With Eosinophilic Duodenitis: Pilot Study
Brief Title: Effectiveness of Biofeedback-Assisted Relaxation Training in Children With Eosinophilic Duodenitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Jennifer Verrill Schurman, Ph.D./Principal Investigator, Children's Mercy Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00003103
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Abdominal Pain; Duodenitis
Keywords: Biofeedback
MeSH Terms: conditions — Abdominal Pain; Duodenitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMT (Active Comparator): Standard Medication Treatment
  Interventions: Behavioral: Biofeedback-assisted relaxation training
- BART (Experimental): Biofeedback-assisted Relaxation Training plus SMT
  Interventions: Behavioral: Biofeedback-assisted relaxation training

INTERVENTIONS:
Behavioral: Biofeedback-assisted relaxation training — 10 sessions BART

SUMMARY:
The purpose of this study is to determine whether the addition of Biofeedback-Assisted Relaxation to standard medication treatment improves outcomes for children with a specific type of recurrent abdominal pain (i.e., eosinophilic gastroenteritis).

DETAILED DESCRIPTION:
Recurrent abdominal pain (RAP) is the most common type of pain in school age children and young adolescents. Previous studies suggest that stress plays an important role in the activation of specific cells that can produce pain within the stomach and intestines. Medication is the standard approach to the treatment of RAP in children. Although medication is helpful for many children, medication alone is not always enough. Biofeedback trains individuals to use relaxation strategies effectively to relieve emotional and physical symptoms, and has been used successfully for stress and pain reduction with both children and adults. It has shown promising results when used alone in the treatment of children with RAP. Research is needed, however, to determine whether biofeedback training is helpful when used in conjunction with medication. Information about how biofeedback training affects the central nervous system and the cells that produce pain also would be useful in refining treatments for this large group of children. The current research will be done in three steps, with Phase 1 designed to evaluate the time, resources, technical support, and sample size needed for successful completion of the full research study. Twenty children (ages 8-18) with eosinophilic duodenitis, a specific form of RAP, will be enrolled and randomly assigned to one of two groups: 1) Standard of Care; or 2) Biofeedback (standard medical care plus 10 sessions of biofeedback training). Measures of pain, functional disability, quality of life, physiological arousal, and global treatment response will be collected pre- and post-intervention, as well as 3 and 6 months later. Data collected will be used to determine how many participants will be needed for the full research study. If biofeedback training is ultimately found to be a positive addition to standard medical treatment, this could lead to improved health outcomes for children with RAP. This information also could result in greater treatment efficiency and reduced health care costs for families, insurance providers, and the hospital system.

ELIGIBILITY:
Inclusion Criteria:

* A current diagnosis of eosinophilic duodenitis per biopsy.
* Ability to participate in the biofeedback training protocol.
* Transportation available to attend twice weekly visits to Children's Mercy Hospital (CMH).

Exclusion Criteria:

* Previous biofeedback training.
* Previous failure of medications used as standard of care in this study.
* Allergy to medications prescribed in this study.
* Co-morbid chronic illness requiring regular medical care.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Primary outcomes involve the feasibility of the method (e.g., compliance with daily diary, salivary cortisol collection) | Up to 6 months

SECONDARY OUTCOMES:
Functional disability rating scale at 6 weeks, 3 months, and 6 months | 6 weeks, 3 months, and 6 months
Pain ratings on daily diary, at 6 weeks, 3 months, and 6 months | 6 weeks, 3 months, and 6 months
Changes in salivary cortisol at 6 weeks, 3 months, and 6 months | 6 weeks, 3 months, and 6 months
Changes in other psychosocial measures (e.g., Behavior Assessment System for Children (BASC), sleep survey, quality of life, etc.) at 6 weeks, 3 months, and 6 months | 6 weeks, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer V Schurman, Ph.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States